CLINICAL TRIAL: NCT02038270
Title: Evolution of the Accuracy of the Nexfin Pressure Signal Compared to Invasive and Noninvasive Arterial Blood Pressure
Brief Title: Accuracy of Nexfin® and NIBP to Predict IBP
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: Nexfin_002
Record Dates: First submitted 2013-05-23; First posted 2014-01-16 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Bloodpressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- surgical patients: 120 Adult patients, that are having a routine surgical procedure.

SUMMARY:
The Nexfin monitoring device relies on noninvasive pressure measurement using a finger-cuff manometer, combined with NIRS technology. The accuracy of the signal is dependent on the degree of vascular unloading, which takes an period before optimal unloading is reached. The evolution of the degree of inaccuracy caused by inclomplete unloading is quantified, and the absolute and relative inaccuracy of the nexfin as a function of the time is determined compared to the invasive blood pressure (IBP).

Secondly, the accuracy of the Nexfin to predict the IBP is compared with the accuracy of noninvasive blood pressure to predict the IBP.

DETAILED DESCRIPTION:
In patients under stable anesthesia conditions, who have IBP and NIBP monitoring, the Nexfin will additionaly be connected. All data will be recorded for at least 30 minutes. NIBP will be measured every 5 minutes The evolution of the NIBP, IBP and Nexfin-derived blood pressure will be analysed to determine the evolution of inaccuracy due to incomplete vascular unloading and to determine the accuracy of Nexfin compared with NIBP to determine IBP.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are accepted for surgery

Exclusion Criteria:

* Patients unable or unwilling to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 Adult patients, that are having a routine surgical procedure.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
vascular unloading time | Start till end of operation
  time to optimal vascular unloading

SECONDARY OUTCOMES:
Bloodpressure | Start till end of operation
  accuracy of nexfin compared to NIBP and IBP

CONTACTS AND LOCATIONS:
Overall Officials: Alain Kalmar, dr, Principal Investigator — univertsity medical center groningen,university of groningen,the netherlands
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands